CLINICAL TRIAL: NCT01816308
Title: Mild Cognitive Impairment (MCI) in Patients With Atrial Fibrillation (AF), Trajectories of the Progression of MCI and Factors Associated With the Progression
Brief Title: Cognitive Impairment in Atrial Fibrillation
Acronym: DIAL-F
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: TCAI_DIAL-F
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation; Mild Cognitive Impairment; Dementia
Keywords: AF; MCI
MeSH Terms: conditions — Atrial Fibrillation; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to compare the incidence of new-onset cognitive impairments and change in existing impairment status between AF patients undergoing either catheter ablation or remaining on anti-arrhythmic drugs (AAD) as assessed by Montreal Cognitive Assessment (MoCA).

DETAILED DESCRIPTION:
Background: AF is mostly a disease of elderly. Up to 10% of people aged 80 years or older suffer from this arrhythmia and the rate is projected to triple in the next 20 years (1). Evidence is emerging that AF may increase the risk of all forms of dementia (2). Cerebral hypoperfusion and the risk of cerebrovascular micro- and macro-embolism are plausible explanations for the predisposition for cognitive decline in AF (1). Such insults may act alone or in concert with other neuropathological changes common in the brain of older individuals such as neuritic plaques or neurofibrillary tangles, in lowering cognitive reserves and accelerating the onset of dementia (3).

Prior studies on AF and dementia have yielded conflicting results.

An earlier study provided evidence supporting an association between AF and increased incidence of dementia in patients with stroke (4). In a prospective study conducted on participants of ONTARGET and TRANSCEND trials, it was revealed that cognitive and functional decline are important consequences of atrial fibrillation, even in the absence of overt stroke (5). Another independent study, observed similar results for risk of dementia in AF in participants with and without clinically recognized stroke during follow-up (3). Evidences from a previous research demonstrated not only a significant association of AF with all forms of dementia including Alzheimer's disease, but also higher mortality rate in patients with coexistent dementia and AF (2). On the contrary, some studies did not find any significant risk-association between AF and dementia (6-8).

These contradictory results compel the necessity for a prospective study on a large population to obtain a clear understanding of the association between AF and cognitive impairment. The potential association between the two conditions can have a very important clinical implication; if there were a causal relationship between AF and dementia then the different therapeutic strategies of AF may have differing influence on dementia risk (3). Thus, this knowledge would facilitate in personalizing treatment approaches for individuals with AF.

Anti-arrhythmic drugs are considered as the first line of therapy in AF and catheter ablation is widely-recognized as the best option in drug-refractory cases. Recent published data suggested that effective rhythm-control by catheter ablation reverses the risk of dementia in AF (9). However, it was an epidemiologic study from a health-care database where ICD codes were used to identify clinical dementia. Therefore, mischaracterization of the dementia subtypes was a major possibility in their study.

None of the other currently ongoing studies or registries on AF ablation in US includes dementia as one of the outcomes to be assessed. Therefore, our study will be the first to examine the benefit of successful catheter ablation on cognitive function in AF patients by directly assessing cognition using standardized instruments.

There are several standardized screening tools available to assess cognitive status, namely Mini-Mental State Examination (MMSE), Cognitive Abilities Screening Instrument (CASI) and Montreal cognitive assessment (MoCA). All have their strengths and limitations, but MoCA is considered the most efficient because of its cross-cultural applicability and its higher sensitivity for detecting mild cognitive impairments. In our study, MoCA would be used to evaluate cognitive status in AF patients.

Besides MoCA, the following questionnaires will be used to assess other risk-factors for cognitive impairment and quality of life in AF patients

1. Hospital anxiety and Depression scale (HAD): to evaluate anxiety and depression
2. Katz Index of Independence in Activities of Daily Living (ADL) and Lawton's Instrumental Activities Of Daily Living Scale (IADL): to assess independent living skills
3. Multidimensional Scale of Perceived Social Support by Zimet et al: to appraise perception of social-support in this study
4. International Physical Activity Questionnaire (IPAQ): to obtain internationally comparable data on health-related physical activity
5. Atrial Fibrillation Effect on Quality-of-Life (AFEQT) questionnaire: to assess the AF-specific changes in QoL before and after ablation

Study Objectives

Primary Objectives:

To evaluate the number of patients showing improvement or no-worsening in cognitive status at 2 years follow-up after catheter ablation or after the beginning of drug-therapy in non-ablation group

Secondary Objectives:

1. Study the interaction between depression, social support and cognitive status
2. Evaluate the impact of social supports on the trajectory of dementia
3. Examine the correlation between physical activity and cognitive impairment
4. Assess the impact of arrhythmia recurrence on dementia across the control and the study group

Study Design:

This prospective multicenter study will enroll 888 consecutive AF patients at different centers in US, Asia and Europe.

Consenting patients will perform the MoCA evaluation. Patients with a score < 17 will be deemed a screen failure. Qualifying patients will be evaluated and the appropriate treatment strategy for managing arrhythmia will be independently determined by the treating physician. Patients undergoing a clinically indicated catheter ablation for AF will be assigned to the Ablation group and those determined to stay on AAD will form the AAD group. Based on physician decision, left atrial appendage occlusion or exclusion procedures may be performed for reducing the thromboembolic risk. The AAD group will continue on AADs as prescribed in accordance with standard of care at the discretion of the physician.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 50 years, male or female subjects
2. Clinical diagnosis of AF
3. Ability to provide written, informed consent

Exclusion Criteria:

1. Patients with established dementia
2. MoCA score ≤ 17 on Montreal Cognitive Assessment (MoCA)
3. Use of illicit drugs
4. Alcohol use: >12 drinks/week on average
5. Clinical evidence of delirium or altered mental status
6. Medically unstable patients (acute/unstable or poorly controlled problems that would demand focused, relatively urgent or emergent medical attention)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Detail study information will be provided to the patients and written informed consent will be obtained from the each patient or family member before enrolling in the study. Consenting patients will be evaluated and the appropriate treatment strategy for managing arrhythmia will be independently determined by the physicians at the participating centers. Patients undergoing catheter ablation for AF will be included in the study group and those determined to stay on AAD will form the control group.
Sampling Method: Non-Probability Sample
Enrollment: 888 (Estimated)
Dates: Start 2014-07; Primary Completion 2020-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
improvement or no-worsening in MoCA score assessed at baseline and 2 year follow-up | 2 years
  The primary efficacy endpoint of this study will be the objective response rate (ORR); objective response being defined as improvement or no-worsening in MoCA score assessed at baseline and 2 year follow-up.

SECONDARY OUTCOMES:
Correlation between MoCA score and physical activity, social support, anxiety and depression | 2 years
  1. Correlation of scores between the HAD and the social support scale
  2. Correlation of scores between HAD and MoCA
  3. Association between social support and MoCA score
  4. Correlation between physical activity and MoCA scale
  5. Association between arrhythmia recurrence and MoCA score
  6. Comparison of QoL between baseline and post-ablation period

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — TCAI; Mitra Mohanty, MD, Study Director — TCAI
Locations (1):
- Texas Cardiac Arrhythmia Institute, St. david's Medical Center, Austin, Texas, United States

REFERENCES:
- [Derived] Mohanty S, Mohanty P, Trivedi C, Assadourian J, Mayedo AQ, MacDonald B, Della Rocca DG, Gianni C, Horton R, Al-Ahmad A, Bassiouny M, Burkhardt JD, Di Biase L, Gurol ME, Natale A. Impact of Oral Anticoagulation Therapy Versus Left Atrial Appendage Occlusion on Cognitive Function and Quality of Life in Patients With Atrial Fibrillation. J Am Heart Assoc. 2021 May 4;10(9):e019664. doi: 10.1161/JAHA.120.019664. Epub 2021 Apr 19. PMID 33870705